CLINICAL TRIAL: NCT04538872
Title: Learning Strategies for Improving Dual Task Performance in Multiple Sclerosis
Acronym: StraDiMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: National MS Center Melsbroek (Other); Revalidatie & MS Centrum Overpelt (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: StraDiMS-001
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MS group implicit (Experimental)
  Interventions: Behavioral: StraDiMS implicit
- MS group explicit (Experimental)
  Interventions: Behavioral: StraDiMs explicit
- HC group implicit (Healthy Controls) (Active Comparator)
  Interventions: Behavioral: StraDiMS implicit
- HC group explicit (Healthy controls) (Active Comparator)
  Interventions: Behavioral: StraDiMs explicit

INTERVENTIONS:
Behavioral: StraDiMS implicit — participants perform a goal-directed stepping task and try to react as fast as possible by stepping on a tile that lights up. Response time (the time between the tile lighting up and the participant stepping on the tile) is the outcome measure of the task. The implicit learning conditions and the explicit learning condition differ from each other in the instructions given prior to the task. The latter group will get more knowledge on the task than the former.
  Arms: HC group implicit (Healthy Controls); MS group implicit
Behavioral: StraDiMs explicit — participants perform a goal-directed stepping task and try to react as fast as possible by stepping on a tile that lights up. Response time (the time between the tile lighting up and the participant stepping on the tile) is the outcome measure of the task. The implicit learning conditions and the explicit learning condition differ from each other in the instructions given prior to the task. The latter group will get more knowledge on the task than the former.
  Arms: HC group explicit (Healthy controls); MS group explicit

SUMMARY:
This study is a randomized controlled study in which we aim to include 60 persons with Multiple Sclerosis and 30 healthy controls. Two different learning strategies, an explicit and an implicit one, will be compared on effects on dual task performance. Further, clinical profile associated with these effects, and brain activity measured by functional near-infrared spectroscopy during dual tasking will be investigated.

To this end, the study will cover 4 days:

Day 1: examine clinical profile; Day 2: baseline dual task measures; Day 3: experimental learning paradigm with subjects randomly assigned to either the implicit or the explicit learning condition.

Day 4: delayed retention dual task and fNIRS measures.

ELIGIBILITY:
Inclusion Criteria:

* all participants: minimal cognitive function (MoCA ≥ 26)
* Persons with MS:

  * Diagnosis of MS
  * EDSS 2.0 - 5.5
  * No relapse within the past 30 days.
  * Able to walk minimally 6 minutes consecutively and to step over the stepping platform without aid.

Exclusion Criteria:

* Other medical conditions interfering with mobility.
* Other neurological conditions.
* Not able to understand instructions.
* Major (unresolvable) problems with hearing or vision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Dual task (STEP + substraction sevens) | day 2
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they continuously subtract sevens, starting from a 3-digit given start number. Duration of the task depends on the speed of the participant (42 steps).
Dual task (STEP + substraction sevens) | day 4
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they continuously subtract sevens, starting from a 3-digit given start number. Duration of the task depends on the speed of the participant (42 steps).
Dual task (STEP + phonetic word list generation) | day 2
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they try to come up with as many words as possible starting with a given letter. Duration of the task depends on the speed of the participant (42 steps).
Dual task (STEP + phonetic word list generation) | day 4
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they try to come up with as many words as possible starting with a given letter. Duration of the task depends on the speed of the participant (42 steps).
Dual task (STEP + Auditory vigilance) | day 2
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they hear a string of letters (1 every 2.5 seconds) and are asked to respond as quickly as possible when they hear the target letter 'L' or 'R'. Duration of the task depends on the speed of the participant (42 steps).
Dual task (STEP + Auditory vigilance) | day 4
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. Concurrently, they will perform a cognitive task in which they hear a string of letters (1 every 2.5 seconds) and are asked to respond as quickly as possible when they hear the target letter 'L' or 'R'. Duration of the task depends on the speed of the participant (42 steps).
Dual Task (WALK + Subtraction sevens) | day 2
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they continuously subtract sevens, starting from a 3-digit given start number. Duration of the task is 30 seconds.
Dual Task (WALK + Subtraction sevens) | day 4
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they continuously subtract sevens, starting from a 3-digit given start number. Duration of the task is 30 seconds.
Dual Task (WALK + Word list generation (phonetic) | day 2
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they try to come up with as many words as possible starting with a given letter. Duration of the task is 30 seconds.
Dual Task (WALK + Word list generation (phonetic) | day 4
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they try to come up with as many words as possible starting with a given letter. Duration of the task is 30 seconds.
Dual Task (WALK + Auditory vigilance) | day 2
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they hear a string of letters (1 every 2.5 seconds) and are asked to respond as quickly as possible when they hear the target letter 'L' or 'R'. Duration of the task is 30 seconds.
Dual Task (WALK + Auditory vigilance) | day 4
  participants will walk on their comfortable, preferred walking speed on a 30-meter walkway. Concurrently, they will perform a cognitive task in which they hear a string of letters (1 every 2.5 seconds) and are asked to respond as quickly as possible when they hear the target letter 'L' or 'R'. Duration of the task is 30 seconds.
learning measure | Day 3
  participants will step as fast as possible on a tile that lights up in a goal-directed stepping task on a platform consisting of 21 stepping tiles. The outcome measure on this task is response time (time from the moment the tile lights up, until the participant steps on the tile).
fNIRS measure (functional near-infrared spectroscopy) | day 4
  a block-design test with 3 tasks (cognitive ST, motor ST and DT) of 25 seconds per task-block (repeated 5 times) will be conducted with a functional near-infrared spectroscopy (fNIRS) neuroimaging system to measure hemoglobin changes during performance of the task and compared between single task and dual task conditions and between groups. Besides, fNIRS will be used during 1 task related to the learning-paradigm.

SECONDARY OUTCOMES:
Age | day 1
height | day 1
weight | day 1
educational level questionnaire | day 1
date of diagnosis questionnaire | day 1
type of MS questionnaire | day 1
EDSS | day 1
  Expanded Disability Status Scale (EDSS)
Digit span forwards visually | day 1
Brief Visuospatial Memory Test (BVMT) | day 1
10/36 Spatial Recall test (SPART) | day 1
Symbol Digit Modalities Test (SDMT) | day 1
Paced Auditory Serial Addition Test (PASAT)-3 seconds | day 1
Digit Span backwards auditory | day 1
6 minute walking test (6MWT) | day 1
Timed-Up and Go (TUG) | day 1
Timed 25 Foot Walk (T25FW) | day 1
4 square stepping test (FSST) | day 1
Berg Balance Scale (BBS) | day 1
Tandem Walk 3m | day 1
Motricity Index | day 1
Movement specific reinvestment scale (MSRS) | day 1
MS Neuropsychological screening questionnaire (MSNQ) | day 1
Multiple Sclerosis Walking Scale (MSWS-12) | day 1
Modified fatigue impact scale (MFIS) | day 1
Activities-specific Balance Confidence scale (ABC) | day 1
Dual Task Questionnaire (DTQ) | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Peter Feys, prof. dr., Principal Investigator — Hasselt University; Renee Veldkamp, drs., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - Noorderhart, Overpelt
  - National MS Center Melsbroek, Steenokkerzeel